CLINICAL TRIAL: NCT03276442
Title: Biological Rhythms in Metabolic Tissues: Impact of Diet
Brief Title: Biorhythms in Metabolic Tissues
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CircHFJC2017
Record Dates: First submitted 2017-08-28; First posted 2017-09-08 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Sleep Deprivation; Metabolic Disturbance; Biological Clocks; Healthy
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Participants will be studied in a crossover design both after a "healthy diet", and after an "unhealthy diet"
Masking Description: In the crossover subgroup condition, participants will not be briefed about what diet they will receive before the actual onset of the dietary intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy diet (Experimental): 'Low-fat dietary intervention' to be administered to participants
  Interventions: Other: Low-fat dietary intervention
- Unhealthy diet (Experimental): 'High-fat dietary intervention' to be administered to participants
  Interventions: Other: High-fat dietary intervention

INTERVENTIONS:
Other: Low-fat dietary intervention — Low-fat diet (5-7 days) preceding extended wakefulness under standardized conditions
  Arms: Healthy diet
Other: High-fat dietary intervention — High-fat diet (5-7 days) preceding extended wakefulness under standardized conditions
  Arms: Unhealthy diet

SUMMARY:
Metabolism is increasingly recognized as being highly regulated by anticipatory biological rhythms (circadian rhythms or "biorhythms"), which are driven by molecular feedback loops, and which are approximately 24 hours long ("circa diem"). These circadian rhythms exist both centrally, in the brain, but also in the periphery, and are specific to many tissues depending on their main biological function or functions. Whereas these circadian rhythms have been thoroughly characterized in other organisms, their role in humans remain poorly understood, partly because of the difficulty in studying these rhythms in peripheral tissues. The investigators therefore aim to characterize these rhythms in primarily skeletal muscle and adipose tissue in healthy young volunteers (using the so-called constant routine paradigm), and how these rhythms interact with one another at various genetic and molecular levels. At the same time, the investigators aim to study how an unhealthy vs. healthy diet can alter these circadian rhythms, and how they interact with circadian rhythms in other tissue compartments such as those expressed by blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-33 yr
* Healthy (self-reported) and not on medication
* BMI 18-28 kg/m2 (and waist circumference <102 cm), and weight stable (±5% body weight in past 6 months)
* Non-smoker and non-nicotine user
* Regular sleep-wake pattern, with sleep duration of 7-9.25 hrs per night
* Sedentary to moderately active with regular exercise habits the last 2 months
* Regular daily meal pattern with 3 main meals

Exclusion Criteria:

* Major or chronic illness, e.g. diabetes, renal disease or inflammatory bowel disease
* Current or history of endocrine or metabolic disorders
* Psychiatric or neurological disorders (e.g. bipolar disorder, epilepsy)
* Frequent gastrointestinal symptoms
* Chronic medication
* Any sleep disorder (e.g. irregular bedtimes, symptoms of insomnia)
* Any issues with or allergies against the provided food items or utilized anesthesia
* Shift work in the preceding three months or for a long duration
* Time travel over two time zones in the preceding month
* Too much weight gain or weight loss in the preceding 6 months
* Pregnancy

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in clock gene & associated omic circadian rhythms | Measured repeatedly (every 6 hours for 24 hours) during a period of extended wakefulness, following each dietary intervention (i.e. over a total period of 6-7 weeks)
  Changes in clock gene & associated clock-regulated & clock-independent metabolic and omic circadian rhythms (e.g. in epigenome, transcriptome, metabolites) in peripheral tissues (primarily skeletal muscle and adipose tissue), and interplay between these rhythms across the 24-h period and under the different dietary conditions

SECONDARY OUTCOMES:
Wakefulness-induced changes and subsequent recovery at omic levels | Following each dietary intervention (i.e. over a total period of 6-7 weeks), measured repeatedly (every 2-6 hours for 24 hours) during a period of extended wakefulness, and after recovery sleep
  Changes at omic levels (e.g. DNA methylation, transcriptome, proteome, metabolome) in peripheral tissues (primarily skeletal muscle and adipose tissue), urine and feces samples due to extended wakefulness following subsequent recovery, following each dietary intervention
24-h rhythms in blood | Measured repeatedly (every 2-3 hours over 24 hours) during a period of extended wakefulness and after subsequent recovery, following each dietary intervention (i.e. over a total period of 6-7 weeks)
  Changes in rhythms in blood-borne cells, proteins and other molecular factors such as DNA, hormones, and proteins, due to the preceding dietary intervention, and relation to other rhythms measured across 24 hrs following the two dietary conditions
Diet-induced changes in gut microbiota and relation to circadian rhythms | Measured throughout study participation, i.e. on average over 6-7 weeks
  Changes in gut microbiota (metagenomic, compositional) due to dietary intervention, and relation to circadian rhythms measured across 24 hrs in peripheral tissues following the two dietary conditions
Energy expenditure rhythms | Measured repeatedly (every 2 hours over 24 hours) during a period of extended wakefulness and after subsequent recovery, following each dietary intervention (i.e. over a total period of 6-7 weeks)
  Changes in energy expenditure rhythms due to the preceding dietary intervention, and relation to other rhythms measured across 24 hrs following the two dietary conditions
Urine metabolite rhythms | Measured throughout study participation, i.e. on average over 6-7 weeks
  Changes in levels of urine metabolites due to dietary intervention, and relation to circadian rhythms across 24 hrs in peripheral tissues following the two dietary conditions
Rhythms of blood markers of damage to the central nervous system | Measured repeatedly (every 1-3 hours over 24 hours) during a period of extended wakefulness and after subsequent recovery, following each dietary intervention (i.e. over a total period of 6-7 weeks)
  Assessment of rhythms in of blood markers of damage to the central nervous system (e.g. Olink Proseek multiplex panel, neuron-specific enolase, S-100b) across a 24-h period and following subsequent recovery sleep, following the two dietary conditions
24-h rhythms in saliva | Measured repeatedly (every 2-3 hours over 24 hours) during a period of extended wakefulness and after subsequent recovery, following each dietary intervention (i.e. over a total period of 6-7 weeks)
  Changes in rhythms in saliva-borne cells, proteins and other molecular factors such as DNA, hormones, and proteins, due to the preceding dietary intervention, and relation to other rhythms measured across 24 hrs following the two dietary conditions
Central circadian rhythms | Measured repeatedly (every 1-3 hours over 24 hours) during a period of extended wakefulness and after subsequent recovery, following each dietary intervention (i.e. over a total period of 6-7 weeks)
  Changes in centrally driven circadian rhythms (e.g. temperature and melatonin), due to the preceding dietary intervention, and relation to other rhythms measured across 24 hrs following the two dietary conditions

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cedernaes, Principal Investigator — Uppsala University
Locations (1):
- Department of Neuroscience, Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brandao LEM, Popa A, Cedernaes E, Cedernaes C, Lampola L, Cedernaes J. Exposure to a more unhealthy diet impacts sleep microstructure during normal sleep and recovery sleep: A randomized trial. Obesity (Silver Spring). 2023 Jul;31(7):1755-1766. doi: 10.1002/oby.23787. Epub 2023 May 28. PMID 37245331